CLINICAL TRIAL: NCT03023007
Title: Study Evaluating the Efficacy of Loco-regional Anaesthesia PECS on the Rate of Chronic Pains 6 Month After a Mastectomy Associated or Not With Axillary Node Dissection and/or a Reconstruction Prosthesis.
Brief Title: Study Evaluating the Efficacy of Loco-regional Anaesthesia PECS on Chronic Pain of a Mastectomy
Acronym: PECS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PECS-1601; N°IdRCB : N°2016-A00562-49 (Other: ANSM)
Record Dates: First submitted 2017-01-10; First posted 2017-01-18 (Estimated); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Breastcancer; Mastectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Loco-regional anaesthesia (Experimental): Loco-regional anaesthesia Anesthesia technique used : loco-regional PECS for patients requiring Mastectomy; And/or Axillary node dissection ; And/or Reconstruction of breast by prosthesis
  Interventions: Procedure: Loco-regional anaesthesia

INTERVENTIONS:
Procedure: Loco-regional anaesthesia — Loco-regional anaesthesia

SUMMARY:
A non-randomized, mono-centric, prospective interventional study that will assess the efficacy of the loco-regional anesthesia PECS on the rate of chronic pain, 6 month after a patient will have either received a mastectomy or a mastectomy associated with axillary nodes dissection, and/or a reconstruction by prosthesis.

DETAILED DESCRIPTION:
The aim of this study is to assess the care given to treat breast cancer while the patient receives a total mastectomy. It is done by evaluating the technique of anesthesia PECS used during this procedure so that the rate of chronic pain can be measured 6 month after the operation.

As well as total mastectomy, patients are also eligible for an axillary lymph node dissection (ALND) and a reconstruction of the breast by prosthesis as options.

Other objectives of the study include:

* Evaluating the effectiveness of the PECS anesthesia technique on the trajectory of acute post-operative pain and on chronic pain after 12 month of the surgery
* Evaluating the type and intensity of the pain
* Evaluating the quality of life
* Study the link between chronic pain and the trajectory of acute pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral breast cancer
* Surgery must be a total mastectomy +/- axillary lymph node dissection and +/- reconstruction by prosthesis; unless first surgery was performed more than 5 years prior to total mastectomy without any residual pain
* Age ≥ 18 ans
* Non-opposition of patients

Exclusion Criteria:

* Reconstruction by other than prosthesis
* Previous breast surgery in the last year
* Hypersensitivity or allergy of anaesthetics
* Coagulopathy and local infections
* Pregnant or breastfeeding
* Patients under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-08-22 (Actual)

PRIMARY OUTCOMES:
Rate of chronic pain | 6 month after surgery
  The rate of chronic pain will be assessed in percentage (%) based on the criteria of the International Association for the Study Pain (IASP) during an algology medical consultation.

SECONDARY OUTCOMES:
Acute post-operative pain | During the 3 days following the surgery
  A representation of the trajectory of pain in the 3 days will be drawn. This pain trajectory is defined as the kinetics of the average daily visual analog scale (VAS) score for 3 days.
Side effects post-operative | During the 3 days following the surgery
  All side effects (e.g. nausea, vomiting etc.) will be recorded, with its date, time, severity, relation with the treatment, treatment associated and evolution. The intensity of adverse events will be scored using the criteria from NCI-CTCAE version 4.0.
Rate of chronic pain | 12 month after the surgery
  Assessed based on the criteria of the International Association for the Study Pain (IASP) collected via telephone call.
Type of chronic pain | 6 and 12 month after surgery
  The type of chronic pain will be determined using the DN4 score. The DN4 score is a form used for the diagnostic of neuropathic pain.
Intensity of chronic pain | 6 and 12 month after surgery
  The intensity of the pain will be recorded using the visual analog scale (VAS).
predictive factors of survival | an average of 1 year
  Using the proportional hazards model.
Quality of life of the patient assessed with the QLQ-C30 questionnaire | an average of 1 year
  QLQ-C30 from the EORTC (quality of life in general, physical condition, limitations to activities, cognitive functions, emotional and social and symptoms occurrences related to cancer or the treatment)
Quality of life of the patient assessed with the QLQ-BR23 questionnaire | an average of 1 year
  QLQ-BR23 (body image, perception of the future etc. and side effects)
Depression assessed with the HADS questionnaire | an average of 1 year
  HADS (Hospital Anxiety and Depression Scale) : to detect anxiety and depression

OTHER OUTCOMES:
Prediction of the post-operative chronic pain with Kalkman score | within the 15 days before the surgery
  The Kalkman score is a validated risk scale based on patient's history and the type of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Abesse AHMEIDI, MD, Study Director — Département Anesthésie /Algologie, Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia V, Wallet J, Leroux-Bromberg N, Delbrouck D, Hannebicque K, Ben Oune F, Leguillette C, Le Deley MC, Ahmeidi A. Incidence and characteristics of chronic postsurgical pain at 6 months after total mastectomy under pectoserratus and interpectoral plane block combined with general anesthesia: a prospective cohort study. Reg Anesth Pain Med. 2024 Jan 11;49(1):36-40. doi: 10.1136/rapm-2022-104185. PMID 37280082